CLINICAL TRIAL: NCT05288023
Title: Azithromycine Pour la Vie Des Enfants au Niger - Implémentation et Recherche: Essai mortalité et résistance (Azithromycin for Child Survival in Niger: Programmatic Trial)
Brief Title: Azithromycin for Child Survival in Niger: Programmatic Trial (AVENIR)
Acronym: AVENIR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: AVENIR I demonstrated efficacy of azithromycin MDA targeted to children 1-59 over 1-11 months in July 2023, thus this trial was stopped before outcomes were collected so Niger could expand the program nationally to include children 1-59 months.
Sponsor: University of California, San Francisco (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Ministry of Health, Niger (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-28387C
Record Dates: First submitted 2022-02-23; First posted 2022-03-18 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Resistance Bacterial; Morality; Child Health; Implementation
MeSH Terms: interventions — Azithromycin; Suspensions

STUDY DESIGN:
Intervention Model Description: Cluster-randomized trial with response adaptive allocation
Masking Description: Participants, investigators, and program implementers will not be actively masked from the study arm allocation given that no placebo will be used. Outcome assessors and data analysts will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Programmatic azithro 1-11 (Active Comparator): Biannual oral azithromycin administration to children aged 1-11 months distributed by community health workers
  Interventions: Drug: Azithromycin for Oral Suspension
- no intervention (No Intervention): No additional intervention.

INTERVENTIONS:
Drug: Azithromycin for Oral Suspension — Azithromycin will be administered as a single dose in oral suspension form for children (up to the maximum adult dose of 1g).
  Dosage will be calculated by age for children aged 1-5 months. For children 6-59 months of age, height-based dosing will be used via height-stick approximation as currently performed by Niger's trachoma program.
  Other Names: Zithromax
  Arms: Programmatic azithro 1-11

SUMMARY:
The MORDOR trial found that biannual distribution of azithromycin to children 1-59 months old reduced child mortality. The World Health Organization (WHO) released conditional guidelines for this intervention, which include targeting azithromycin distributions to children 1-11 months of age in high mortality settings. The proposed trial aims to demonstrate and evaluate large-scale implementation of azithromycin to children aged 1-11 months old in the context of a programmatic setting while monitoring mortality and resistance antimicrobial resistance.

DETAILED DESCRIPTION:
In the Programmatic Trial, community health centers (also known as "CSIs" or "Centres de Santé Intégrés") will be randomized to one of two arms: 1) programmatic azithro 1-11: biannual oral azithromycin administration to children aged 1-11 months distributed by community health workers or 2) no intervention: no distribution of azithromycin. A total of 2,490 communities within selected CSIs will be included .

All communities in both arms receive routine health services offered by community health workers working for the Niger Ministry of Health's community health program.

Mortality will be monitored through birth histories. Mortality and morbidity will also be monitored using routinely collected community and clinic visit data. Antimicrobial resistance will be monitored in a subset of eligible CSIs.

ELIGIBILITY:
Intervention

At the community-level, eligibility includes:

Inclusion Criteria:

* Location in Dosso, Tahoua, Maradi, Zinder, or Tillabéri regions
* Distinguishable from neighboring communities
* Verbal consent of community leader(s)

Exclusion criteria:

* Inaccessible or unsafe for study team
* "Quartier" designation on national census

At the individual-level, eligibility includes:

Inclusion criteria:

* Age 1-11 months
* Primary residence in a study community
* Verbal consent of caregiver/guardian for study participation

Exclusion criteria:

* Known allergy to macrolides

Population-based sample collections

At the community-level, eligibility includes:

Inclusion criteria:

* Location in study region
* Distinguishable from neighboring communities
* Verbal consent of community leader(s)

Exclusion criteria:

* Inaccessible or unsafe for study team
* Included in MORDOR trials
* Not randomly selected

At the individual-level, eligibility includes:

Inclusion criteria:

* Age 1-59 months or 7-12 years or caregiver/guardian of a child eligible for treatment
* Primary residence in a study community selected for sample collections
* Verbal consent of caregiver/guardian for study participation

Exclusion criteria:

* Not on list of randomly selected participants from the census

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 169707 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kieran O'Brien, PhD, MPH, Principal Investigator — University of California, San Francisco; Tom Lietman, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Proctor foundation, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data underlying outcomes publications will be made publicly available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual participant data will be made available after publication of the outcomes and will be made available indefinitely.
Access Criteria: Once made available, the data will be open access.

REFERENCES:
- [Background] WHO Guideline on Mass Drug Administration of Azithromycin to Children under Five Years of Age to Promote Child Survival [Internet]. Geneva: World Health Organization; 2020. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK561641/ PMID 32924384
- [Background] Keenan JD, Bailey RL, West SK, Arzika AM, Hart J, Weaver J, Kalua K, Mrango Z, Ray KJ, Cook C, Lebas E, O'Brien KS, Emerson PM, Porco TC, Lietman TM; MORDOR Study Group. Azithromycin to Reduce Childhood Mortality in Sub-Saharan Africa. N Engl J Med. 2018 Apr 26;378(17):1583-1592. doi: 10.1056/NEJMoa1715474. PMID 29694816

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Health Center
Groups:
- Programmatic Azithro 1-11: Biannual oral azithromycin administration to children aged 1-11 months distributed by community health workers
  Azithromycin for Oral Suspension: Azithromycin will be administered as a single dose in oral suspension form for children (up to the maximum adult dose of 1g).
  Dosage will be calculated by age for children aged 1-5 months. For children 6-59 months of age, height-based dosing will be used via height-stick approximation as currently performed by Niger's trachoma program.
Period: Overall Study
Arm/Group | Programmatic Azithro 1-11 | no Intervention
Started | 135754; 110 Health Center | 33953; 56 Health Center
Completed | 135754; 110 Health Center | 33953; 56 Health Center
Not Completed | 0; 0 Health Center | 0; 0 Health Center

BASELINE CHARACTERISTICS:
Population: Inclusion criteria includes: age 1-59 months, primary residence in a study community, verbal consent of caregiver/guardian of children for study participation, weight ≥ 3.0 kg.
  Children were enrolled for participation. not guardians.
  The No Intervention arm data was not collected given the pragmatic design of the trial; therefore, the Programmatic Azithro 1-11 data was used to estimate the No Intervention population (33,953).
Groups:
- Total: Total of all reporting groups
Arm/Group | Programmatic Azithro 1-11 | No Intervention | Total
Number analyzed (Participants) | 135,754 | 33,953 | 169707
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 135,754 | 33,953 | 169707
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex was not recorded
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Niger | 135,754 | 33,953 | 169707

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Genetic Determinants of Macrolide Resistance From Population-based Samples
Description: Prevalence of genetic determinants of macrolide resistance including those determinants known to be found in Streptococcus pneumoniae, Streptococcus pyogenes, and Staphylococcus aureus in nasopharyngeal swabs in children aged 1-59 months from population-based samples after 1 year of distribution
Time Frame: 2 years
Population: The study stopped prior to the collection of outcome measures.
Arm/Group | Programmatic Azithro 1-11 | no Intervention
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Load of Genetic Determinants of Macrolide Resistance From Population-based Samples
Description: Load of genetic determinants of resistance to macrolides including those determinants known to be found in Campylobacter spp, Salmonella spp, Shigella spp, and Escherichia coli from rectal swabs in children 1-59 months old from population-based samples, defined as read number per million base pairs, using DNA-seq (metagenomic deep sequencing).
Time Frame: 2 years
Population: The study stopped prior to the collection of outcome measures.
Arm/Group | Programmatic Azithro 1-11 | no Intervention
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Prevalence of Genetic Determinants of Macrolide Resistance From Clinic-based Samples
Description: Prevalence of resistance to macrolides including those determinants known to be found in Streptococcus pneumoniae, Streptococcus pyogenes, and Staphylococcus aureus from nasopharyngeal swabs in children 1-59 months old.
Time Frame: 2 years
Population: The study stopped prior to the collection of outcome measures.
Arm/Group | Programmatic Azithro 1-11 | no Intervention
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Load of Genetic Determinants of Macrolide Resistance From Clinic-based Samples
Description: Load of genetic determinants of resistance to macrolides including those determinants known to be found in Campylobacter spp, Salmonella spp, Shigella spp, and Escherichia coli from rectal swabs in children 1-59 months old, defined as read number per million base pairs, using DNA-seq (metagenomic deep sequencing).
Time Frame: 2 years
Population: The study stopped prior to the collection of outcome measures.
Arm/Group | Programmatic Azithro 1-11 | no Intervention
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of All-cause Clinic Visits
Description: Number of all-cause clinic visits per month for children aged 1-59 months over 1 year
Time Frame: 2 years
Population: The study stopped prior to the collection of outcome measures.
Arm/Group | Programmatic Azithro 1-11 | no Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Reporting adverse event data began with the first round of treatment through the last round of treatment. If a child experiences an adverse event within 28 days of treatment, it was reported. time frame for reporting was 12 months
Description: According to Pfizer, a serious adverse event (SAE) is any adverse event that: results in death, Is life-threatening (i.e., causes an immediate risk of death), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity. Or that is considered to be: an important medical event.
Arm/Group | Programmatic Azithro 1-11 | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/135754 | 0/33953
Serious Adverse Events (participants affected / at risk) | 0/135754 | 0/33953
Other Adverse Events (participants affected / at risk) | 0/135754 | 0/33953

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT05288023/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT05288023/SAP_001.pdf